CLINICAL TRIAL: NCT02078401
Title: Ophthalmological Screening and Follow-up of Optic Pathway Gliomas in Children With Neurofibromatosis Type 1.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Catherine Cassiman, MD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S56406
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Neurofibromatosis Type 1
Keywords: Optic pathway glioma; Ophthalmological screening
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neurofibromatosis type 1 children

SUMMARY:
The goal of this project is to get more insight into the (neuro)ophthalmological characteristics of children with neurofibromatosis type 1. This way investigators would like to update the current guidelines for follow up and treatment of optic pathway gliomas. Clinical findings will be compared with the results of Optical coherence tomography (OCT) and MRI (magnetic resonance imaging).

ELIGIBILITY:
Inclusion Criteria:

* neurofibromatosis type 1

Exclusion Criteria:

* no neurofibromatosis type 1

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with neurofibromatosis type 1 with and without optic pathway glioma
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | childhood (0 to 18y)
Presence of optic pathway glioma | childhood (0 to18y)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cassiman, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium